CLINICAL TRIAL: NCT03491670
Title: Iron Metabolism After Out of Hospital Cardiac Arrest
Brief Title: Free Iron and Out of Hospital Cardiac Arrest
Acronym: DESFER
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DESFER (29BRC17.0154)
Record Dates: First submitted 2018-03-26; First posted 2018-04-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2019-11

CONDITIONS: Arrest Cardio Respiratory
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Out of hospital cardiac arrest is associated with a poor prognosis. The aim of this study is to provide a better understanding of perturbations of iron metabolism after cardiac arrest and to analyze the impact on clinical centered outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to ICU for out of hospital cardiac arrest
* Therapeutic hypothermia

Exclusion Criteria:

* Absence of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU for out of hospital cardiac arrest
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 year
  Mortality

SECONDARY OUTCOMES:
Neurologic outcome | 6 months post cardiac arrest
  Cerebral Performance Categories scale, ranging from 1 to 5, with a patient considered "1" when he has good cerebral performance and 5 when he has very poor cerebral performance (including brain death)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the international committee of Brest UH. Requestors will be required to sign and completet a data access agreement